CLINICAL TRIAL: NCT04757142
Title: PLASMA Chile (PLASMA Chile)
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT20035
Record Dates: First submitted 2021-02-03; First posted 2021-02-17 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multicenter, observational cohort study to collect data on Chilean patients diagnosed with Heart Failure with reduced ejection fraction, their treatments, and their progress in a real-world environment. Additional objectives will be analyzed, such as mortality, and the barriers, if any, to receiving the indicated treatment.

DETAILED DESCRIPTION:
Identify the main epidemiological and clinical characteristics of patients with Heart Failure with reduced ejection fraction, as well as the medical treatment models used.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years old.
* Patients with Heart Failure with Left Ventricular Ejection Fraction (LVEF) ≤ 40% will be included.
* Patients must be willing to comply with the study requirements and complete the Informed Consent Form (defined as the legally valid and documented confirmation of a patient's voluntary agreement to participate in the clinical study).

Exclusion Criteria:

* Patients without Heart Failure or with Heart Failure with Left Ventricular Ejection Fraction (LVEF)> 40%.
* Patients unable to comply with the Clinical Investigation Plan.
* Patients who are already enrolled or plan to participate in a concurrent clinical study of any medication and/or device at any time during the course of this clinical study without prior documented approval of the Medtronic Study Manager.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chilean patients diagnosed with Heart Failure with reduced ejection fraction, regardless of the time of disease progression.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Identify the main epidemiological and clinical characteristics of patients with Heart Failure with reduced ejection fraction, as well as the medical treatment models used. | 1 year
  Patient´s baseline characteristics, medical history, socio-economic data, ancillary studies, laboratory tests, and cardiovascular medication will be summarized using summary statistics. Continuous variables will be presented using mean, standard deviation (SD), minimum, median, maximum, and interquartile range (IQR). Categorical variables will be presented as frequency and percentage.

SECONDARY OUTCOMES:
Determine the prescription rate of a cardiovascular pharmacological treatment in patients with Heart Failure with reduced ejection fraction | 1 year
  Percentage of cardiovascular medication prescription by type
Determine the prescription rate of a cardiac medical device in patients with Heart Failure with reduced ejection fraction | 1 year
  Percentage of patients with an indication for a cardiac medical device.
Determine the implant rate of a cardiac medical device in patients with Heart Failure with reduced ejection fraction | 1 year
  Percentage of patients implanted with a cardiac medical device.
Determine the mortality rate and its classification in patients with Heart Failure with reduced ejection fraction during a 12-month period. | 1 year
  Percentage of deaths during the study follow-up period Number and percentage of deaths according to their classification. Risk assessment of sudden cardiac death in the population. Risks comparison of sudden death at 6 and 12 months of follow-up
Determine the hospitalization rate for heart failure during the 12-month follow-up. | 1 year
  Percentage of Hospitalizations during the study follow-up period.
Identify the barriers, if any, to prescribing and implanting a cardiac medical device in those patients with a Class I recommendation according to the ACC/AHA/HRS 2017 guidelines. | 1 year
  Percentage of reasons for not indicating a cardiac medical device. Number and percentage of reasons for not implanting a cardiac medical device
Determine the population with a profile of 1.5 primary prevention of sudden cardiac death | 1 year
  Frequency of patients with indication for 1.5 primary prevention of sudden cardiac death (patients with Heart Failure in primary prevention who have one or more of the following risk factors: syncope or pre-syncope; left ventricular ejection fraction less than 25%; presence of non-sustained ventricular tachycardia; more than 10 ventricular extrasystoles per hour observed in a 24-hour Holter)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Muratore, MD, Study Director — Medtronic
Locations (6):
- Chile (6):
  - Hospital Clínico Regional Guillermo Grant Benavente, Concepción
  - Hospital Clínico Pontificia Universidad Católica de Chile, Santiago
  - Hospital San Juan de Dios, Santiago
  - Hospital Talagante, Santiago
  - Hospital Hernan Henriquez Aravena, Temuco
  - Hospital Dr. Gustavo Fricke, Viña del Mar

IPD SHARING:
Plan to Share IPD: No